CLINICAL TRIAL: NCT06384339
Title: ID-ClimAct. Influence of Social Motives of Clients and Staff on the Social Climate of Secure Settings
Acronym: ID-ClimAct
Status: Completed | Type: Observational
Sponsor: University Psychiatric Clinics Basel (Network)
Collaborators: University of Basel (Other)
Responsible Party: Principal Investigator, Andrea Canel, Principal Investigator, University Psychiatric Clinics Basel
Other Study IDs: ID-ClimAct-1
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Social Environment; Correctional Institutions; Rehabilitation of Criminals; Social Dominance; Interpersonal Relations
MeSH Terms: conditions — Social Dominance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clients: Adult clients in a secure setting (i.e. prison or forensic mental health psychiatry
  Interventions: Diagnostic Test: CSIV, Social motive; Diagnostic Test: Interpersonal messages and behavior; Diagnostic Test: CCS, Social motive
- Staff: Adult staff in a secure setting (including forensic healthcare staff, social workers, probation officers, prison offers, education staff)
  Interventions: Diagnostic Test: CSIV, Social motive; Diagnostic Test: Interpersonal messages and behavior; Diagnostic Test: CCS, Social motive

INTERVENTIONS:
Diagnostic Test: CSIV, Social motive — The CSIV is a self-report measure and assesses interpersonal values using eight octant scales, which are aggregated into overall communion and agency scores, ranging from -4 to +4 .
  Other Names: Circumplex Scales of Interpersonal Values (CSIV; Locke, 2000)
Diagnostic Test: Interpersonal messages and behavior — The Impact Message Inventory - Circumplex (IMI-C) Brief Version is a self-report transactional inventory designed to measure a target person's interpersonal behavior on four octant scales dominance, hostility, submissiveness, and friendliness by assessing the covert responses or "impact messages" of another person. Each subscale consists of 7 items, with each item scored on a 4-point Likert scale from 1 (not at all) to 4 (very much so). The minimum score per scale is 7 and the maximum score is 28.
  Other Names: Impact Message Inventory - Circumplex (IMI-C; Kiesler, 2006)
Diagnostic Test: CCS, Social motive — The CCS is a elf-report inventory, that measures tendencies towards competitiveness versus caring in social interactions. The minimum score for the two subscales competitiveness and caring are 9 and the maximum score is 90.
  Other Names: Competitiveness and Caring Scale (CCS; McEwan, Gilbert, & Duarte, 2012)

SUMMARY:
The social climate in secure settings is an essential element to successful rehabilitation. Previous studies indicate that staff characteristics are a relevant factor contributing to a beneficial social climate. Yet, secure settings form a specific and challenging work environment. Staff members are faced with clients who present a variety of difficult emotional and behavioural problems. Social motives for caring and cooperation can be blocked in a threatening environment, favouring dysfunctional interpersonal dynamics between individuals. This observational study explores the reciprocal influences of social motives between clients and staff on the social climate within secure settings.

ELIGIBILITY:
Inclusion Criteria:

* Clients who are currently incarcerated within the specified secure settings.
* Staff members currently employed in the specified secure settings.
* Individuals (both clients and staff) who are capable of providing informed consent.
* Clients who are deemed competent and not under any disciplinary restrictions that would preclude participation.
* Staff members who are directly involved with client care and management.

Exclusion Criteria:

* Clients who are not considered competent to provide informed consent.
* Staff members who do not have direct interactions with clients (e.g., administrative staff not involved in direct care).
* Clients and staff from open prisons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will involve approximately 200 participants, consisting of both clients and staff members from various secure settings such as prisons and forensic psychiatries in Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Social Climate Perception | Day 1
  Measured through Essen Climate Evaluation Schema (EssenCES). The EssenCES uses a 5-point Likert scale for each item, ranging from 0 (never) to 4 (always). The three subscales Therapeutic Hold, Patients' Cohesion and Experienced Safety each comprises five items, the minimum score for each subscale is 0 and the maximum is 20.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Graf, Prof. Dr., Study Director — University Psychiatric Clinics Basel
Locations (1):
- University Psychiatric Clinics Basel, Clinic for Forensics, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No